CLINICAL TRIAL: NCT06481111
Title: Prospective Monocentric Registry of Patients Undergoing Vitamin D Treatment at San Raffaele Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Di Filippo, Medical Physician Specialist in Endocrinology, IRCCS San Raffaele
Other Study IDs: "REGIDO"
Record Dates: First submitted 2024-06-04; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: supplementary treatment with vitamin D — observational design

SUMMARY:
The Endocrinology Unit of the IRCCS San Raffaele Hospital is dedicated to establishing a prospective single-center registry with data from patients undergoing vitamin D supplementation, initiating their first visit to the outpatient unit until December 2029. 1000 patients will be enrolled, aligning with the unit's recent patient influx for hypovitaminosis D.

The registry's goal is to assess the epidemiological trend, identify risk factors, and evaluate the diagnostic and therapeutic clinical management strategies for hypovitaminosis D. It will involve collecting clinical, laboratory, and historical data during outpatient visits, adhering to the standard diagnostic and therapeutic protocols for endocrine-metabolic diseases. This data collection is expected to continue for a duration of ten years.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (age ≥ 18 years) regardless of fertility status and pregnancy/breastfeeding conditions
* Vitamin D supplementation, with any formulation and dosage
* Signing of informed consent

Exclusion Criteria:

* Patients unable to understand and sign informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatient clinics who will access of the Endocrinology Unit of the IRCCS San Raffaele Hospital for endocrine-metabolic diseases and who are on supplementary treatment with vitamin D until December 2029
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of data in outpatient accessing Endocrinology Unit of the IRCCS San Raffaele Hospital for endocrine-metabolic diseases who are on supplementary treatment with vitamin D. | 10 years
  The main outcome of the study is to assess the prevalence changes of major comorbidities and their complications including cardiovascular diseases, diabetes, cancer, and osteoporosis, during the study-period in relation to the use and characteristics of vitamin D supplementation, in order to evaluate the potential influence of vitamin D use on patient's outcomes. The pathological conditions will be diagnosed according to current major guidelines and clinical practice.

IPD SHARING:
Plan to Share IPD: No